CLINICAL TRIAL: NCT07322250
Title: The Effect of Blood Flow Restriction Training on Postmenopausal Stress Urinary Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Hamdiah Mohmmed Altuwjry, physical therapist, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-800
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Post Menopausal Stress Urinary Incontinence
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Control group will receive Pelvic floor muscle training-associated EMG biofeedback.
  Interventions: Other: pelvic floor muscle training -associated EMG-biofeedback.
- experimental group (Experimental): experimental group will receive Pelvic floor muscle training-associated EMG biofeedback while applying blood flow restriction to the proximal thigh.
  Interventions: Other: pelvic floor muscle training -associated EMG-biofeedback.; Other: blood flow restriction

INTERVENTIONS:
Other: pelvic floor muscle training -associated EMG-biofeedback. — The control group will receive pelvic floor muscle training-associated EMG biofeedback for 10 weeks
Other: blood flow restriction — experimental group will receive Pelvic floor muscle training-associated EMG biofeedback while applying blood flow restriction to the proximal thigh for 10 weeks.
  Arms: experimental group

SUMMARY:
the purpose of the study is to investigate the effect of blood flow restriction training on postmenopausal SUI.

DETAILED DESCRIPTION:
We have two groups: control group (A) and experimental group (B) are two matched post-menopausal stress urinary incontinence. Group A will receive PFMT-associated EMG biofeedback, whereas Group B will receive PFMT-associated EMG biofeedback while applying blood flow restriction to the proximal thigh. Our primary outcome measures will be the severity of SUI symptoms, while the secondary outcome measures will involve QOL, self-esteem, patient's global impression of improvement, maximum voluntary isometric contraction (MVIC) of pelvic floor muscles, pelvic floor muscle resting tone, and the endurance of pelvic floor muscles,

ELIGIBILITY:
Inclusion Criteria:

1. post-menopausal women, defined by the absence of vaginal bleeding for 12 months,
2. body mass index (BMI) < 30
3. They should have faced at least two leakage episodes each week and fall into the mild to moderate range of urinary incontinence, measured by (ICIQ-UI SF).
4. Two standard questions about stress and urgency UI were used to determine the patient's eligibility.

Exclusion Criteria:

1. pelvic organ prolapse greater than grade II on Baden-Walker classification system
2. previous treatment for UI or hormone therapy, ongoing urinary tract infections, cognitive or neurological disorder, or inability to perform the proposed procedures.
3. anyone with past or current injuries to the pelvis, hip joint, or spine, as well as those with uncontrolled diabetes, or those with prior experience in pelvic floor muscle training .
4. the presence of uncontrolled hypertension.
5. patients with a history of deep venous thrombosis (DVT), varicose Veins, cardiac disease, or lymphedema.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
severity of stress urinary incontinence (SUI) symptoms. | baseline,10 weeks, 16 weeks
  severity of SUI symptoms, measured by the Arabic version of the International consultation on incontinence questionnaire-short form (ICIQ-UI SF)

SECONDARY OUTCOMES:
Quality of life (QOL) | baseline,10 weeks, 16 weeks
  QOL will be measured by International consultation on incontinence questionnaire Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTS qol)
self-esteem | baseline,10 weeks, 16 weeks
  self-esteem will be measured by Arabic Rosenberg self-esteem scale
patient's global impression of improvement | baseline,10 weeks, 16 weeks
  patient's global impression of improvement will be measured by Patient Global Impression of Improvement (PGI-I) scale.
maximum voluntary isometric contraction (MVIC) of pelvic floor muscles | baseline,10 weeks, 16 weeks
  maximum voluntary isometric contraction (MVIC) of pelvic floor muscles will be measured by Neurotrac myoplus pro EMG
pelvic floor muscle resting tone | baseline,10 weeks, 16 weeks
  pelvic floor muscle resting tone will be measured by Neurotrac myoplus pro EMG
pelvic floor muscle endurance | baseline,10 weeks, 16 weeks
  pelvic floor muscle endurance will be measured by Neurotrac myoplus pro EMG